CLINICAL TRIAL: NCT02589548
Title: Brazilian Prospective Hodgkin Lymphoma Registry
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Responsible Party: Principal Investigator, Irene Biasoli, Associate Professor, Universidade Federal do Rio de Janeiro
Other Study IDs: RBLH
Record Dates: First submitted 2015-10-26; First posted 2015-10-28 (Estimated); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Hodgkin Lymphoma; Hodgkin Disease
Keywords: Hodgkin Lymphoma; Hodgkin Disease
MeSH Terms: conditions — Hodgkin Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Formalin-fixed tissue for central diagnostic pathology review
Oversight: Data Monitoring Committee: No

SUMMARY:
The study is a prospective registry of Hodgkin Lymphoma (HL) patients in Brazil.

The purpose of the study is to gather clinical, epidemiologic and outcomes data on the treatment of HL, on the basis of records collected by key Brazilian institutions, through a centralized web-based registry of clinical data verified by central board of hematopathologists.

DETAILED DESCRIPTION:
Hodgkin Lymphoma is considered one of the malignancies with highest cure rates. Its prognosis improved substantially along the last three decades, as a result of relevant cooperative studies carried out in American and European institutions. Around 70-80% of the patients are cured with the available chemotherapy regimens.

However, data about HL in developing countries are scarce. It is well established that patients in underprivileged societies present with malignancies in more advanced stages. In studies of HL patients treated in Brazil during the 80's, most patients presented with advanced disease.

The creation of registry of patients with HL will provide a more reliable picture of the disease in the country, its prevalence in different areas and socioeconomic groups, and treatment outcomes. It will also foster the establishment of a network among hospitals in all regions of the country, which may serve as a platform for further development of cooperative studies engaging the main Brazilian Institutions.

The data collection allows comparison of data entered into the registry against predefined rules for range or consistency with other data fields in the registry. Also, quality assurance addresses data validation and data analysis. Standard descriptive analyses will be carried out. For a crude association analysis, categorical data will be analysed using the chi-square or Fisher's exact test (two-sided). Survival curves will be estimated using the Kaplan-Meier method and compare using the log-rank test. Univariate and multivariate Cox regression analyses will be conducted to verify the prognostic factors regarding Progression free survival and Overall survival, adjusted for relevant prognostic clinical variables and treatment.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated HL patients
* Clinical data including baseline information on disease localization and laboratory parameters at staging, features of treatment adopted and assurance of follow-up updating for at least 5 years are requested
* Written informed consent

Exclusion Criteria:

-

Ages: 12 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hodgkin Lymphoma patients
Sampling Method: Non-Probability Sample
Enrollment: 1400 (Estimated)
Dates: Start 2009-10; Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 5 years
  Overall Survival

SECONDARY OUTCOMES:
Event Free survival | 5 years
  Event free survival

CONTACTS AND LOCATIONS:
Overall Officials: Nelson Spector, MD, Study Chair — UFRJ; Irene Biasoli, Principal Investigator — UFRJ
Locations (1):
- Universidade Federal Do Rio de Janeiro, Rio de Janeiro, Brazil